CLINICAL TRIAL: NCT03921177
Title: Micronutrient Supplementation Before and During 1st Pregnancy to Improve Birth Outcomes (JiVitA-5)
Acronym: JiVitA-5
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Extended COVID-19 restrictions on field research and limited funding
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: JiVitA Project, Gaibandha, Bangladesh (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB 7841
Record Dates: First submitted 2019-04-11; First posted 2019-04-19 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Birth Weight; Miscarriage; Small-for-gestational Age; Preterm Birth
Keywords: preconceptional multiple micronutrient supplementation; periconceptional multiple micronutrient supplementation; pregnancy outcomes; adolescent pregnancy; Bangladesh
MeSH Terms: conditions — Birth Weight; Abortion, Spontaneous; Premature Birth

STUDY DESIGN:
Intervention Model Description: Cluster-randomized, placebo-controlled concurrent intervention trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Multiple micronutrient and placebo tablets are identical in size, shape, and appearance; coding of supplements carried out independent of investigators and research team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiple micronutrient supplement (Experimental): Daily micronutrient supplement
  Interventions: Dietary Supplement: Multiple micronutrient supplement
- Placebo (Placebo Comparator): Daily identifcal placebo tablet
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Dietary Supplement: Multiple micronutrient supplement — Preconception to 12-weeks gestation: daily (coded) multiple micronutrient supplement containing 15-nutrients (vitamins and minerals) providing an approximate recommended dietary allowance for pregnant women, approximating the UNICEF UNIMAP formulation (UN micronutrient preparation).
  Arms: Multiple micronutrient supplement
Drug: Placebo Oral Tablet — Preconception to 12-weeks gestation: identical tablet
  Arms: Placebo

SUMMARY:
The purpose of this cluster-randomized trial is to evaluate the efficacy of daily, multiple micronutrient (MM) supplement versus identical placebo use among nulligravid, recently married women, starting preconceptionally through the 1st trimester of pregnancy, in reducing low birth weight and other adverse pregnancy outcomes in rural Bangladesh.

DETAILED DESCRIPTION:
Micronutrient deficiencies are common among women of reproductive age in rural South Asia, including Bangladesh. Antenatal multiple micronutrient (MM) supplementation, usually starting toward the end of the 1st trimester, has been shown to reduce low birth weight in many cultures. In northern Bangladesh, where the current study will be conducted, MM versus iron-folic acid supplementation has been shown to extend gestational age, thereby reducing risks of preterm birth 15% and low birth weight by 12%, and reduce risk of stillbirth by 11% (West KP et al. JAMA 2014), and to reduce risk of micronutrient deficiencies (Schulze KJ et al J Nutr 2019). Since it is plausible that women of reproductive age conceive in a state of lower micronutrient nutriture, it remains unknown the degree to which MM supplementation, starting preconceptionally through the 1st trimester (covering the periconceptional and embryonic period) can benefit pregnancy outcome. Further, there is concern that newlywed, nulligravid women in rural South Asia are at high risk, and may be at particular health and pregnancy risks due to micronutrient deficiencies resulting from dietary inadequacy.

The investigators propose to conduct a double-masked, cluster-randomized, placebo-controlled trial among recently married women in 18 rural unions of Gaibandha District, Bangladesh, that will provide a daily tablet containing either (a) a MM formulation containing a US Institute of Medicine (IOM) Recommended Dietary Allowance (RDA) for pregnancy for 15 essential vitamins and minerals (and closely approximates the UNIMAP formula), or (b) a placebo tablet of identical appearance containing no micronutrients, during a period extending from at least one-month prior to last menstrual period through the 1st trimester of pregnancy (~12 weeks' gestation). The study area will comprise 566 rural clusters (sectors) each with 250-400 households, serving as units of randomization. Consenting, recently married women will be detected through routine community surveillance and start to receive coded, double-masked supplements, resupplied during monthly home visits. Participating women will receive coded supplements for daily consumption until the end of the trial or until determined to be pregnant. On detection of pregnancy by a history of amenorrhea confirmed by urine test, irrespective of randomized allocation, all women will be switched to receive an open-labeled MM supplement, expected to occur toward the end of the 1st trimester, which will continue through 3 months post-partum. This switch is in response to previous positive effects shown on pregnancy outcomes with a MM supplement starting at the end of the 1st trimester.

Participating married women will be periodically interviewed for socioeconomic, morbidity, dietary and lifestyle risk factors and assessed by anthropometry. Pregnancies will be followed for miscarriage, abortion, live birth and still birth outcomes. Newborn anthropometry will be assessed to determine birth weight and size. Infants and mothers will be eligible for additional breast feeding, dietary, morbidity and growth assessments at 8 days, and 1, 3 and 6 months after delivery. Participating women resident in a predefined subset of the study area (n~68 sectors) will receive enhanced assessments, including blood draw in the end of the 1st trimester for subsequent laboratory assessment of micronutrient status, and body composition, among other measures.

ELIGIBILITY:
Inclusion Criteria:

* Resident of 566 rural sectors (clusters) in Gaibandha district
* Recently-married woman
* Nulligravid

Exclusion Criteria:

* Women with a history of previous pregnancy
* Women who refuse consent for participation

Max Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 9859 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-05-29 (Actual)

PRIMARY OUTCOMES:
Preterm Birth - number of live-births occurring earlier than 37 weeks gestation among all live-births (with known gestational age) | up to 38 weeks of gestation
  Pregnancies ending in a live birth less than 37 weeks' gestation
Miscarriage - number of spontaneous abortions occurring earlier than 24 weeks gestation among all pregnancies (with known gestational age) | up to 24 weeks gestation
  Pregnancies ending as a spontaneous abortion less than 24 weeks' gestation
Small for Gestational Age - number of live-born neonates weighing less than the 10th centile of birth weight for gestational age and sex among all live-births (with known gestational age and birth weight) | up to 72 hours after live birth
  Infants weighing less than the 10th centile of birth weight for gestational age and sex
Low Birth Weight - number of live-born neonates weighing less than 2500 g at birth among all live-births (with known birth weight) | Measured from time of live birth through 72 hours after birth
  Infants weighing less than 2500 g at birth

SECONDARY OUTCOMES:
Anemia in Pregnant Women | Measured at 12 weeks gestation
  Hemoglobin in whole blood, less than a cutoff of 110 g/L
Iron Status | Measured at 12 weeks gestation
  Distribution of plasma ferritin, ng/mL
Vitamin A Status | Measured at 12 weeks gestation
  Distribution of plasma retinol, micromoles/L
Vitamin E Status | Measured at 12 weeks gestation
  Distribution of plasma alpha-tocopherol, micromoles/L
Folate Status | Measured at 12 weeks gestation
  Distribution of total plasma folate, nmol/L
Vitamin B12 Status | Measured at 12 weeks gestation
  Distribution of total plasma cobalamin, pmol/L
Selenium Status | Measured at 12 weeks gestation
  Distribution of total plasma selenium, ng/mL

CONTACTS AND LOCATIONS:
Overall Officials: Keith P West, Jr., DrPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- JiVitA Project Office, Gaibandha, Gaibandha Distict, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
To be delineated
Supporting Information: Study Protocol
Time Frame: Not later than 4 years after completion of data collection in the field
Access Criteria: To be delineated

REFERENCES:
- [Background] West KP Jr, Shamim AA, Mehra S, Labrique AB, Ali H, Shaikh S, Klemm RD, Wu LS, Mitra M, Haque R, Hanif AA, Massie AB, Merrill RD, Schulze KJ, Christian P. Effect of maternal multiple micronutrient vs iron-folic acid supplementation on infant mortality and adverse birth outcomes in rural Bangladesh: the JiVitA-3 randomized trial. JAMA. 2014 Dec 24-31;312(24):2649-58. doi: 10.1001/jama.2014.16819. PMID 25536256
- [Background] Sugimoto JD, Labrique AB, Ahmad S, Rashid M, Klemm RD, Christian P, West KP Jr. Development and management of a geographic information system for health research in a developing-country setting: a case study from Bangladesh. J Health Popul Nutr. 2007 Dec;25(4):436-47. PMID 18402187
- [Background] Gernand AD, Schulze KJ, Stewart CP, West KP Jr, Christian P. Micronutrient deficiencies in pregnancy worldwide: health effects and prevention. Nat Rev Endocrinol. 2016 May;12(5):274-89. doi: 10.1038/nrendo.2016.37. Epub 2016 Apr 1. PMID 27032981
- [Background] Labrique AB, Christian P, Klemm RD, Rashid M, Shamim AA, Massie A, Schulze K, Hackman A, West KP Jr. A cluster-randomized, placebo-controlled, maternal vitamin A or beta-carotene supplementation trial in Bangladesh: design and methods. Trials. 2011 Apr 21;12:102. doi: 10.1186/1745-6215-12-102. PMID 21510905